CLINICAL TRIAL: NCT06208657
Title: Optimal Precision TherapIes to CustoMISE Care in Childhood and Adolescent Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Australian & New Zealand Children's Haematology/Oncology Group (Other)
Collaborators: The Hospital for Sick Children (Other); Medical Research Future Fund (Other); Kazia Therapeutics Limited (Industry); C17 Council (Other); Bristol-Myers Squibb (Industry); Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMISE; ANZCHOG2204 (Other: ANZCHOG)
Record Dates: First submitted 2023-12-12; First posted 2024-01-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Childhood Cancer; Childhood Solid Tumor; Childhood Brain Tumor; Recurrent Cancer; Refractory Cancer
Keywords: children; basket trial; platform study; pediatric; solid tumor; paediatric; solid tumour; CNS tumor; CNS tumour; lymphoma
MeSH Terms: conditions — Neoplasms; Recurrence; Central Nervous System Neoplasms; Lymphoma | interventions — Opdualag; Irinotecan; Pharmaceutical Preparations; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A Paxalisib (Experimental): Drug: Irinotecan, Drug: Temozolomide, Drug: Paxalisib. Irinotecan starting at 50mg/m2/day, intravenous, on days 1-5, 28 day cycle, 13 cycles.
  Temozolomide starting at 150mg/m2/day, oral, on days 1-5, 28 day cycle, 13 cycles.
  Paxalisib starting at 21mg/m2 oral, daily, 28 day cycle, 13 cycles.
  Interventions: Drug: Paxalisib; Drug: Irinotecan (drug); Drug: Temozolomide (TMZ)
- Arm C Opdualag (Experimental): Drug: Opdualag, a fixed dose combination of Nivolumab and Relatlimab Opdualag, a fixed-dose combination of Nivolumab 480mg and Relatlimab 160mg, intravenous, on day 1, 28 day cycle, 26 cycles.
  Interventions: Drug: Opdualag

INTERVENTIONS:
Drug: Paxalisib — Paxalisib starting at 21mg/m2 oral, daily, 28 day cycle, 13 cycles.
  Arms: Arm A Paxalisib
Drug: Opdualag — Opdualag, a fixed-dose combination of Nivolumab 480mg and Relatlimab 160mg, intravenous, on day 1, 28 day cycle, 26 cycles
  Arms: Arm C Opdualag
Drug: Irinotecan (drug) — Irinotecan starting at 50mg/m2/day, intravenous, on days 1-5, 28 day cycle, 13 cycles.
  Arms: Arm A Paxalisib
Drug: Temozolomide (TMZ) — Temozolomide starting at 150mg/m2/day, oral, on days 1-5, 28 day cycle, 13 cycles.
  Arms: Arm A Paxalisib

SUMMARY:
A companion platform trial to test novel targeted agents based on the patient's tumor profile.

DETAILED DESCRIPTION:
Both Australia (Zero Childhood Cancer) and Canada (PROFYLE) have developed precision oncology programs for the pediatric population through which samples from childhood/adolescent cancers undergo in depth genetic profiling. OPTIMISE is a companion platform trial, which will link patients to novel targeted agents based on their tumor profile. The trial will have multiple basket arms based on the most common genetically altered pathways the investigators have identified in these childhood cancers. Each arm of the trial will be histopathology agnostic and test a rational, novel combination therapy, to maximise potential clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with a solid tumor, CNS tumor or lymphoma that has progressed despite standard therapy, or for which no effective standard therapy exists.
2. Age <21 years at inclusion; patients 21 years and older may be included after approval by the Study Chair if they have a pediatric type recurrent/refractory malignancy.
3. Patients must be enrolled on a precision medicine study (i.e. PROFYLE, ZERO or equivalent as agreed with Study Chair).
4. Patients enrolled in a Phase I cohort must have either evaluable or measurable disease.
5. Patients enrolled in a Phase II cohort must have measurable disease. Evaluable and measurable disease are defined by standard imaging criteria for the patient's tumor type.
6. Disease evaluations, laboratory tests, and other clinical assessments that are considered standard of care may be undertaken at the patient's local oncology treatment centre with results transferred to study site for evaluation.
7. Performance status: Karnofsky performance status (for patients > 16 years of age) or Lansky play score (for patients ≤ 16 years of age) ≥ 50%.
8. Life expectancy ≥ 6 weeks.
9. Patients must have fully recovered from the acute toxic effects of all prior anticancer therapy and must meet the following minimum duration from prior anticancer-directed therapy prior to enrolment.
10. Adequate organ function.
11. Able to comply with scheduled follow-up and with management of toxicity.
12. Females of childbearing potential must have a negative serum or urine pregnancy test.
13. Fertile males must agree to use adequate contraception during the study and following completion of treatment.
14. Provide a signed and dated informed consent form.

Exclusion Criteria:

1. Patients with symptomatic central nervous system (CNS) primary or metastatic tumours who are neurologically unstable or require increasing doses of corticosteroids or local CNS-directed therapy to control their CNS disease. Patients on stable doses of corticosteroids for at least 7 days prior to receiving study drug may be included.
2. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, or malabsorption syndrome) - only for arms that include orally administered therapeutic agents.
3. Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality), unstable ischemia, congestive heart failure within 12 months of screening.
4. Known active viral hepatitis or human immunodeficiency virus (HIV) infection or any other uncontrolled infection.
5. Major surgery within 21 days of the first dose of investigational drug. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumour biopsy and insertion of central venous access devices are not considered major surgery, but for these procedures, a 48-hour interval must be maintained before the first dose of the investigational drug is administered.
6. Known hypersensitivity to any study drug or component of the formulation.
7. Pregnant or nursing (lactating) females.
8. Any other concomitant serious medical condition or organ dysfunction that in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the investigational drug(s).

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants treated with molecularly-targeted agents in each treatment arm. | 5 Years
  Number of CAYA participants (children, adolescents and young adults) with advanced solid tumours (including CNS tumors and non-Hodgkin lymphomas) where molecular sequencing data was used to allocate treatment arms of molecularly-targeted agents.
Recommended phase II dose for each treatment arm | 3 Years
  Recommended phase II dose of a novel single agent or combination treatment in CAYA participants, determined by dose-limiting toxicities reported as per CTCAE V5.0.
Objective Response Rate (ORR) for each treatment arm. | 5 Years
  ORR defined as complete response and partial response, as measured by RECIST, RAPNO, INRC or RECIL in CAYA participants treated with molecularly-targeted agents.

SECONDARY OUTCOMES:
Overall Clinical Benefit Rate (CBR) for each treatment arm | 5 Years
  CBR defined as complete response and partial response and stable disease, as measured by RECIST, RAPNO, INRC or RECIL in CAYA participants treated with molecularly-targeted agents.
Progression Free Survival (PFS) for each treatment arm. | 5 Years
  PFS in CAYA participants from initiation of treatment with molecularly-targeted agents to the occurrence of disease progression, as measured by RECIST, RAPNO, INRC or RECIL, or death.
Incidence of treatment-emergent adverse events for each treatment arm. | 5 Years
  Safety and tolerability of molecularly-targeted agents as measured by incidence of treatment-emergent adverse events reported as per CTCAE V5.0 in CAYA participants.
Maximum Concentration (Cmax) of molecularly-targeted agents for each treatment arm. | 5 Years
  Cmax in plasma after the first dose of molecularly-targeted agents in CAYA participants.

CONTACTS AND LOCATIONS:
Overall Officials: David Ziegler, Prof, Study Chair — Sydney Children's Hospital - Australian Study Chair; Daniel Morgenstern, Dr, Study Chair — The Hospital for Sick Children - Canadian Study Chair
Locations (14):
- Australia (9):
  - John Hunter Children's Hospital, Newcastle, New South Wales
  - Sydney Children's Hospital, Randwick, Sydney, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Children's Hospital, Melbourne, Victoria
  - The Royal Children's Hospital, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (5):
  - Stollery Children's Hospital, Edmonton
  - CHU Sainte Justine, Montreal
  - Children's Hospital of Eastern Ontario, Ottawa
  - The Hospital for Sick Children, Toronto
  - BC Children's Hospital, Vancouver

IPD SHARING:
Plan to Share IPD: Yes
Plan to Share IPD: Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the Sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the Study Committee.
  The pseudonymized data will be shared for transparency reasons in the context of publications and after publication with other physicians and scientists (national and international academia) to promote and accelerate research on causes and treatment development of oncological diseases.
  Requests for access to pseudonymized patient data for other scientific purposes will be reviewed by the Study Committee. A positive statement of the respective ethic committee and a signed data protection commitment are requested. Results of scientific research based on the study data may be used for academic teaching, research and scientific publications or presentations at scientific meetings.